CLINICAL TRIAL: NCT01895361
Title: A Phase II, Multicenter, Randomized, Placebo-Controlled, Double-Blind, 12-Month Study to Assess Safety and Efficacy of SelG1 With or Without Hydroxyurea Therapy in Sickle Cell Disease Patients With Sickle Cell-Related Pain Crises
Brief Title: Study to Assess Safety and Impact of SelG1 With or Without Hydroxyurea Therapy in Sickle Cell Disease Patients With Pain Crises
Acronym: SUSTAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Reprixys Pharmaceutical Corporation (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SelG1-00005; R44HL093893 (NIH); R01FD004805 (FDA)
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Sickle Cell Disease
Keywords: SelG1; P-selectin; monoclonal antibody; sickle cell disease; sickle cell anemia; sickle cell; pain crisis; pain crises; vasoocclusion; vaso-occlusion; priapism; hepatic sequestration; splenic sequestration; chest syndrome; SCD
MeSH Terms: conditions — Anemia, Sickle Cell; Priapism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High-dose SelG1 (Selg1 5.0 mg/kg) (Experimental): IV Infusion, once every 4 weeks through Week 50
  Interventions: Drug: SelG1
- Low-dose SelG1 (Selg1 2.5 mg/kg) (Experimental): IV Infusion, once every 4 weeks through Week 50
  Interventions: Drug: SelG1
- Placebo (Placebo Comparator): IV Infusion, once every 4 weeks through Week 50
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SelG1
  Arms: High-dose SelG1 (Selg1 5.0 mg/kg); Low-dose SelG1 (Selg1 2.5 mg/kg)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine whether the investigational drug SelG1 when given to sickle cell disease patients either taking or not taking hydroxyurea was effective in preventing or reducing the occurrence of pain crises. SelG1 prevents various cells in the bloodstream from sticking together. By stopping these cell-cell interactions, SelG1 may prevent small blood vessels from becoming blocked and therefore reduce the occurrence and severity of pain crises. Other effects of SelG1 was evaluated, as well as the safety of the drug and how long it stayed in the blood stream.

Funding Source - FDA Office of Orphan Products Development (OOPD)

ELIGIBILITY:
Key Inclusion Criteria:

* Sickle Cell Disease (HbSS, HbSC, HbSβ⁰-thalassemia, or HbSβ⁺-thalassemia)
* If receiving hydroxyurea or erythropoietin, treatment must have been prescribed for at least 6 months, with the dose stable for at least 3 months
* Between 2 and 10 sickle cell-related pain crises in the past 12 months

Key Exclusion Criteria:

* On a chronic transfusion program or planning on exchange transfusion during the study
* Hemoglobin <4.0 g/dL
* Planned initiation, termination, or dose alteration of hydroxyurea during the study
* Receiving chronic anticoagulation therapy (e.g. warfarin, heparin) other than aspirin

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2013-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (56):
- United States (49):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Little Rock, Arkansas
  - Los Angeles, California
  - Oakland, California
  - Orange, California
  - Sacramento, California
  - Aurora, Colorado
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Daytona Beach, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - Peoria, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Jackson, Mississippi
  - Kansas City, Missouri
  - Las Vegas, Nevada
  - New Brunswick, New Jersey
  - Newark, New Jersey
  - Brooklyn, New York
  - New Hyde Park, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Greenville, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Sumter, South Carolina
  - Fort Worth, Texas
  - Houston, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
- Brazil (6):
  - Salvador, Estado de Bahia
  - Porto Alegre, Rio Grande do Sul
  - Campinas, São Paulo
  - São José Do Rio Preto, São Paulo
  - Rio de Janeiro
  - São Paulo
- Kingston, Jamaica

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Sy SKB, Tanaka C, Grosch K. Population Pharmacokinetics and Pharmacodynamics of Crizanlizumab in Healthy Subjects and Patients with Sickle Cell Disease. Clin Pharmacokinet. 2023 Feb;62(2):249-266. doi: 10.1007/s40262-022-01193-4. Epub 2022 Dec 18. PMID 36529836
- [Derived] Kanter J, Brown RC, Norris C, Nair SM, Kutlar A, Manwani D, Shah N, Tanaka C, Bodla S, Sanchez-Olle G, Albers U, Liles D. Pharmacokinetics, pharmacodynamics, safety, and efficacy of crizanlizumab in patients with sickle cell disease. Blood Adv. 2023 Mar 28;7(6):943-952. doi: 10.1182/bloodadvances.2022008209. PMID 36355805
- [Derived] Ataga KI, Kutlar A, Kanter J, Liles D, Cancado R, Friedrisch J, Guthrie TH, Knight-Madden J, Alvarez OA, Gordeuk VR, Gualandro S, Colella MP, Smith WR, Rollins SA, Stocker JW, Rother RP. Crizanlizumab for the Prevention of Pain Crises in Sickle Cell Disease. N Engl J Med. 2017 Feb 2;376(5):429-439. doi: 10.1056/NEJMoa1611770. Epub 2016 Dec 3. PMID 27959701

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approx. 174 patients were planned. A total of 198 patients were randomized. 192 patients received at least 1 dose of study drug & were analyzed for safety; 198 patients were analyzed for efficacy, 125 patients contributed data to the analysis of SelG1 PK data, & 176 patients contributed data to the analysis of PD data (% P-selectin inhibition).
Pre-assignment Details: The study included a Screening Phase, Treatment Phase, and Follow-up Evaluation Phase. During the Screening Phase, potential study participants were to be fully screened for both inclusion and exclusion criteria before and undergo clinical and laboratory evaluations within 30 days prior to randomization into the study.
Groups:
- High-dose SelG1 (Selg1 5.0 mg/kg); Low-dose SelG1 (Selg1 2.5 mg/kg): IV Infusion, once every 4 weeks through Week 50
  SelG1
- Placebo: IV Infusion, once every 4 weeks through Week 50
  Placebo
Period: Overall Study
Arm/Group | High-dose SelG1 (Selg1 5.0 mg/kg) | Low-dose SelG1 (Selg1 2.5 mg/kg) | Placebo
Started | 67 | 66 | 65
Completed | 43 | 45 | 41
Not Completed | 24 | 21 | 24
Not completed — Adverse Event | 1 | 1 | 3
Not completed — Death | 2 | 1 | 2
Not completed — Lost to Follow-up | 4 | 4 | 6
Not completed — Non-compliance with study | 1 | 3 | 1
Not completed — Physician Decision | 2 | 2 | 2
Not completed — Withdrawal by Subject | 7 | 6 | 6
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Reasons different from categories above | 7 | 3 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT): The ITT population includes all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | High-dose SelG1 (Selg1 5.0 mg/kg) | Low-dose SelG1 (Selg1 2.5 mg/kg) | Placebo | Total
Number analyzed (Participants) | 67 | 66 | 65 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (10.89) | 30.1 (9.79) | 29.3 (10.36) | 30.1 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 38 | 109
  Male | 32 | 30 | 27 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 12 | 11 | 43
  Not Hispanic or Latino | 45 | 52 | 53 | 150
  Unknown or Not Reported | 2 | 2 | 1 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 60 | 62 | 60 | 182
  White | 4 | 2 | 3 | 9
  Other | 3 | 2 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Annual Rate of Sickle Cell-related Pain Crises (SCPC) Per Hodges-Lehmann Median
Description: An SCPC is defined as an acute episode of pain with no other medically determined cause than a vasoocclusive event that requires a medical facility visit and treatment with oral or parenteral narcotics, or parenteral non-steroidal anti-inflammatory drugs. The annual rate of SCPC is defined as the total number of pain crises for a patient occurring from the date of randomization to the end date multiplied by 365 divided by the number of days during that same time period. End date is defined as the last dose date plus 14 days. For participants never dosed, the end date was the end of study date. This calculation accounts for early dropouts or lost to follow-up by extrapolating the SCPC rate of every participant to one year.
Time Frame: One year
Population: Intent-to-Treat (ITT) population: The ITT population includes all randomized participants.
Measure: Median (Full Range); unit: SCPC per year
Arm/Group | High-dose SelG1 (Selg1 5.0 mg/kg) | Low-dose SelG1 (Selg1 2.5 mg/kg) | Placebo
Number analyzed (Participants) | 67 | 66 | 65
SCPC per year | 1.63 [0.0 to 24.3] | 2.01 [0.0 to 24.3] | 2.98 [0.0 to 24.3]
Statistical Analysis 1: Comparison: High-dose SelG1 (Selg1 5.0 mg/kg) vs Placebo; Test type: Other; p = 0.010, Stratified Wilcoxon Rank Sum Test; with HU therapy (yes, no) and categorized crisis history (2 to 4, 5 to 10) as recorded in the IXRS system as the strata; Hodges-Lehmann median absolute diff. = -1.01, 95% CI 2-sided [-2.00 to 0.00]
Statistical Analysis 2: Comparison: Low-dose SelG1 (Selg1 2.5 mg/kg) vs Placebo; Test type: Other; p = 0.180, Stratified Wilcoxon Rank Sum Test; with HU therapy (yes, no) and categorized crises history (2 to 4, 5 to 10) as recorded in the IXRS system as the strata; Hodges-Lehmann median absolute diff. = -0.69, 95% CI 2-sided [-1.84 to 0.02]

2. Primary Outcome: Annual Rate of Sickle Cell-related Pain Crises (SCPC) - Per Standard Median
Description: as for outcome 1
Time Frame: One year
Population: Intent-to-Treat (ITT) population: The ITT population includes all randomized participants.
Measure: Median (Full Range); unit: SCPC per year
Arm/Group | High-dose SelG1 (Selg1 5.0 mg/kg) | Low-dose SelG1 (Selg1 2.5 mg/kg) | Placebo
Number analyzed (Participants) | 67 | 66 | 65
SCPC per year | 1.63 [0.0 to 24.3] | 2.01 [0.0 to 24.3] | 2.98 [0.0 to 24.3]
Statistical Analysis 1: Comparison: High-dose SelG1 (Selg1 5.0 mg/kg) vs Placebo; Test type: Other; Change vs placebo (%) = -45.3
Statistical Analysis 2: Comparison: Low-dose SelG1 (Selg1 2.5 mg/kg) vs Placebo; Test type: Other; Change vs placebo (%) = -32.6

3. Secondary Outcome: Annual Rate of Days Hospitalized (Key Secondary Endpoint) Per Hodges-Lehmann Median
Description: The annual rate of days hospitalized was calculated as the number of days hospitalized multiplied by 365 divided by the end date minus the date of randomization plus one where the end date is defined as the last dose date plus 14 days (for subjects never dosed, the end date equaled the end of study date, which was the last site contact for these patients).
Time Frame: One year
Population: ITT: The ITT population includes all randomized patients.
Measure: Median (Full Range); unit: Days hospitalized per year
Arm/Group | High-dose SelG1 (Selg1 5.0 mg/kg) | Low-dose SelG1 (Selg1 2.5 mg/kg) | Placebo
Number analyzed (Participants) | 67 | 66 | 65
Days hospitalized per year | 4.00 [0.0 to 130.7] | 6.87 [0.0 to 151.0] | 6.87 [0.0 to 307.4]
Statistical Analysis 1: Comparison: High-dose SelG1 (Selg1 5.0 mg/kg) vs Placebo; Test type: Other; p = 0.450, Stratified Wilcoxon Rank Sum Test; with HU therapy (yes, no) and categorized crises history (2 to 4, 5 to 10) as recorded in the IXRS system as the strata; Hodges-Lehmann median absolute diff. = 0.00, 95% CI 2-sided [-4.36 to 0.00]
Statistical Analysis 2: Comparison: Low-dose SelG1 (Selg1 2.5 mg/kg) vs Placebo; Test type: Other; p = 0.837, Stratified Wilcoxon Rank Sum Test; with HU therapy (yes, no) and categorized crises history (2 to 4, 5 to 10) as recorded in the IXRS system as the strata; Hodges-Lehmann median absolute diff. = 0.00, 95% CI 2-sided [-3.90 to 2.61]

4. Secondary Outcome: Time to First Sickle Cell-related Pain Crisis
Description: Time to first SCPC is defined as months from randomization to first SCPC. A participant without SCPC before withdrawal or completion of the study is considered censored at the time of the end date. End date is defined as the last dose plus 14 days. For participants never dosed, the end date is the end of study date.
Time Frame: Up to one year
Population: ITT population: The ITT population includes all randomized participants.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | High-dose SelG1 (Selg1 5.0 mg/kg) | Low-dose SelG1 (Selg1 2.5 mg/kg) | Placebo
Number analyzed (Participants) | 67 | 66 | 65
months | 4.07 [1.31 to NA] — NA = insufficient number of participants with events | 2.20 [0.95 to 6.60] | 1.38 [0.39 to 4.90]
Statistical Analysis 1: Comparison: High-dose SelG1 (Selg1 5.0 mg/kg) vs Placebo; Test type: Other; p = 0.001, Log Rank; Hazard Ratio (HR) = 0.495, 95% CI 2-sided [0.331 to 0.741] — Calculated based on Cox regression analysis with HU therapy (yes, no), categorized crises history (2 to 4, 5 to 10), and treatment as covariates
Statistical Analysis 2: Comparison: Low-dose SelG1 (Selg1 2.5 mg/kg) vs Placebo; Test type: Other; p = 0.136, Log Rank; Hazard Ratio (HR) = 0.752, 95% CI 2-sided [0.515 to 1.097] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Time to Second Sickle Cell-related Pain Crisis
Description: Time to second SCPC is defined as months from randomization to second SCPC. A patient with less than two SCPC before withdrawal or completion of the study is considered censored at the time of the end date. End date is defined as the last dose plus 14 days. For patients never dosed, the end date is the end of study date.
Time Frame: Up to one year
Population: ITT population: The ITT population includes all randomized participants.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | High-dose SelG1 (Selg1 5.0 mg/kg) | Low-dose SelG1 (Selg1 2.5 mg/kg) | Placebo
Number analyzed (Participants) | 67 | 66 | 65
months | 10.32 [4.47 to NA] — NA = insufficient number of participants with events | 9.20 [3.94 to 12.16] | 5.09 [2.96 to 11.01]
Statistical Analysis 1: Comparison: High-dose SelG1 (Selg1 5.0 mg/kg) vs Placebo; Test type: Other; p = 0.022, Log Rank; Hazard Ratio (HR) = 0.534, 95% CI 2-sided [0.329 to 0.866] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Low-dose SelG1 (Selg1 2.5 mg/kg) vs Placebo; Test type: Other; p = 0.100, Log Rank; Hazard Ratio (HR) = 0.693, 95% CI 2-sided [0.440 to 1.092] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Annual Rate of Uncomplicated Sickle Cell-related Pain Crisis Per Hodges-Lehmann Median
Description: Uncomplicated SCPC is defined as an acute episode of pain with no known cause for pain other than a vasoocclusive event; requiring a visit to a medical facility; and requiring treatment with a parenteral or oral narcotic (including opiates), or parenteral NSAIDs; but is NOT classified as an acute chest syndrome, hepatic sequestration, splenic sequestration or priapism.
Time Frame: Up to one year
Population: ITT population: The ITT population includes all randomized participants.
Measure: Median (Full Range); unit: Uncomplicated SCPC per year
Arm/Group | High-dose SelG1 (Selg1 5.0 mg/kg) | Low-dose SelG1 (Selg1 2.5 mg/kg) | Placebo
Number analyzed (Participants) | 67 | 66 | 65
Uncomplicated SCPC per year | 1.08 [0.0 to 24.3] | 2.00 [0.0 to 24.3] | 2.91 [0.0 to 19.2]
Statistical Analysis 1: Comparison: High-dose SelG1 (Selg1 5.0 mg/kg) vs Placebo; Test type: Other; p = 0.015, Stratified Wilcoxon Rank Sum Test; with HU therapy (yes, no) and categorized crises history (2 to 4, 5 to 10) as recorded in the IXRS system as the strata; Hodges-Lehmann median absolute diff. = -1.00, 95% CI 2-sided [-1.98 to 0.00]
Statistical Analysis 2: Comparison: Low-dose SelG1 (Selg1 2.5 mg/kg) vs Placebo; Test type: Other; p = 0.120, Stratified Wilcoxon Rank Sum Test; with HU therapy (yes, no) and categorized crises history (2 to 4, 5 to 10) as recorded in the IXRS system as the strata; Hodges-Lehmann median absolute diff. = -0.87, 95% CI 2-sided [-1.77 to 0.00]

7. Secondary Outcome: Annual Rate of Acute Chest Syndrome Per Hodges-Lehmann Median
Description: Acute Chest Syndrome (ACS) is defined on the basis of the finding of a new pulmonary infiltrate involving at least one complete lung segment that was consistent with alveolar consolidation, but excluding atelectasis (as indicated by chest X-ray). At least one of the following additional signs or symptoms needs to be present as well: a participant had to have reported chest pain, a temperature of more than 38.5oC, tachypnea, wheezing or cough.
Time Frame: One year
Population: ITT population: The ITT population includes all randomized participants.
Measure: Median (Full Range); unit: accute chest syndrome per year
Arm/Group | High-dose SelG1 (Selg1 5.0 mg/kg) | Low-dose SelG1 (Selg1 2.5 mg/kg) | Placebo
Number analyzed (Participants) | 67 | 66 | 65
accute chest syndrome per year | 0.00 [0.0 to 3.7] | 0.00 [0.0 to 3.9] | 0.00 [0.0 to 24.3]
Statistical Analysis 1: Comparison: High-dose SelG1 (Selg1 5.0 mg/kg) vs Placebo; Test type: Other; p = 0.780, Stratified Wilcoxon Rank Sum test; with HU therapy (yes, no) and categorized crises history (2 to 4, 5 to 10) as recorded in the IXRS system as the strata; Hodges-Lehmann median absolute diff. = 0.00, 95% CI 2-sided [0.00 to 0.00]
Statistical Analysis 2: Comparison: Low-dose SelG1 (Selg1 2.5 mg/kg) vs Placebo; Test type: Other; p = 0.868, Stratified Wilcoxon Rank Sum test; with HU therapy (yes, no) and categorized crises history (2 to 4, 5 to 10) as recorded in the IXRS system as the strata; Hodges-Lehmann median absolute diff. = 0.00, 95% CI 2-sided [0.00 to 0.00]

8. Secondary Outcome: Patient Reported Outcome: Change From Baseline in Pain Severity/Pain Interference Domain From Brief Pain Inventory (BPI) Questionnaire
Description: The BPI instrument was completed by the patients at pre-specified study visits prior to & during the Treatment & Follow-Up Evaluation Phases. Patients completed the brief pain inventory long-form, 1-week recall at the indicated pre-specified study visits. The BPI is a standardized self-reported questionnaire developed to provide information on the intensity of pain (the sensory dimension) as well as the degree to which pain interferes with function (the reactive dimension). The BPI also asks questions about pain relief, pain quality, & the patient's perception of the cause of pain. Since pain can be quite variable over a day, the BPI asks patients to rate their pain at the time of responding to the questionnaire (pain now), & also at its worst, least, & average over the previous week. The scorings for pain & interference have a range from 0 (no pain/no interference) to 10 (worst pain/complete interference). The BPI scoring manual was used to calculate scores for each domain.
Time Frame: Baseline, Day 15, Week 14, Week 26, Week 38, Week 52, and Week 58, up to 58 weeks
Population: ITT population: The ITT population includes all randomized participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High-dose SelG1 (Selg1 5.0 mg/kg) | Low-dose SelG1 (Selg1 2.5 mg/kg) | Placebo
Number analyzed (Participants) | 67 | 66 | 65
score on a scale
  Pain Severity: Baseline (BL) (n=48,49,55): number analyzed (Participants) | 48 | 49 | 55
  Pain Severity: Baseline (BL) (n=48,49,55) | 4.363 (2.1176) | 4.531 (2.0089) | 4.129 (2.0076)
  Pain Severity: CFB to Day 15 (n=38,42,47): number analyzed (Participants) | 38 | 42 | 47
  Pain Severity: CFB to Day 15 (n=38,42,47) | -0.123 (1.3419) | 0.073 (1.5097) | 0.355 (1.7289)
  Pain Severity: CFB to Week (Wk) 14 (n=32,33,33): number analyzed (Participants) | 32 | 33 | 33
  Pain Severity: CFB to Week (Wk) 14 (n=32,33,33) | -0.146 (1.1520) | -0.068 (1.4608) | -0.152 (2.0918)
  Pain Severity: CFB to Week 26 (n=27,31,32): number analyzed (Participants) | 27 | 31 | 32
  Pain Severity: CFB to Week 26 (n=27,31,32) | -0.377 (1.2460) | -0.290 (1.9865) | -0.563 (2.3751)
  Pain Severity: CFB to Week 38 (n=25,29,29): number analyzed (Participants) | 25 | 29 | 29
  Pain Severity: CFB to Week 38 (n=25,29,29) | -0.267 (1.4079) | 0.026 (1.3893) | 0.333 (1.8430)
  Pain Severity: CFB to Week 52 (n=18,23,22): number analyzed (Participants) | 18 | 23 | 22
  Pain Severity: CFB to Week 52 (n=18,23,22) | -0.634 (1.8501) | 0.130 (1.5899) | -0.310 (1.9508)
  Pain Severity: CFB to Wk 58 follow up (n=27,33,30): number analyzed (Participants) | 27 | 33 | 30
  Pain Severity: CFB to Wk 58 follow up (n=27,33,30) | -0.145 (1.2309) | 0.091 (1.3790) | -0.444 (1.8626)
  Pain Interference: BL (n=48,49,55): number analyzed (Participants) | 48 | 49 | 55
  Pain Interference: BL (n=48,49,55) | 4.643 (2.5726) | 4.656 (2.6099) | 4.995 (2.9470)
  Pain Interence: CFB to Day 15 (n=38,42,47): number analyzed (Participants) | 38 | 42 | 47
  Pain Interence: CFB to Day 15 (n=38,42,47) | -0.674 (2.2868) | -0.099 (2.0435) | -0.816 (2.3556)
  Pain Interence: CFB to Wk 14 (n=32,33,33): number analyzed (Participants) | 32 | 33 | 33
  Pain Interence: CFB to Wk 14 (n=32,33,33) | -0.213 (2.3988) | -0.534 (2.7769) | -0.039 (3.0412)
  Pain Interference: CFB to Wk 26 (n=27,32,32): number analyzed (Participants) | 27 | 32 | 32
  Pain Interference: CFB to Wk 26 (n=27,32,32) | -0.583 (2.2844) | -0.728 (2.4220) | -0.821 (3.1561)
  Pain Interference: CFB to Wk 38 (n=25,29,29): number analyzed (Participants) | 25 | 29 | 29
  Pain Interference: CFB to Wk 38 (n=25,29,29) | -0.866 (2.7720) | -0.119 (1.6473) | -0.221 (3.1076)
  Pain Interference: CFB to Wk 52 (n=18,23,22): number analyzed (Participants) | 18 | 23 | 22
  Pain Interference: CFB to Wk 52 (n=18,23,22) | -1.014 (2.0989) | -0.174 (2.2510) | -0.819 (2.8490)
  Pain Interference: CFB to Wk 58 f/up (n=27,33,30): number analyzed (Participants) | 27 | 33 | 30
  Pain Interference: CFB to Wk 58 f/up (n=27,33,30) | -0.476 (2.3473) | -0.386 (2.2249) | -0.802 (2.5785)

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) timeframe: Adverse events were collected from first dose of study treatment until end of study treatment, up to a maximum duration of 58 weeks.
Description: Adverse Event (AE): Any sign or symptom that occurs during the study treatment. Of the 198 patients randomized, 192 received at least one dose of study treatment and were included in the Safety set.
Groups:
- High-dose SelG1 (5.0 mg/kg SelG1); Low-dose SelG1 (2.5 mg/kg SelG10; Placebo: IV Infusion, once every 4 weeks through Week 50
Arm/Group | High-dose SelG1 (5.0 mg/kg SelG1) | Low-dose SelG1 (2.5 mg/kg SelG10 | Placebo
All-Cause Mortality (participants affected / at risk) | 2/66 | 1/64 | 2/62
Serious Adverse Events (participants affected / at risk) | 17/66 | 21/64 | 17/62
Other Adverse Events (participants affected / at risk) | 46/66 | 47/64 | 42/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-dose SelG1 (5.0 mg/kg SelG1) (N=66) | Low-dose SelG1 (2.5 mg/kg SelG10 (N=64) | Placebo (N=62)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 1
BRADYCARDIA (Cardiac disorders) | 1 | 0 | 0
PALPITATIONS (Cardiac disorders) | 0 | 1 | 0
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 0 | 0 | 1
SICKLE CELL ANAEMIA WITH CRISIS (Congenital, familial and genetic disorders) | 1 | 0 | 2
HYPERPARATHYROIDISM PRIMARY (Endocrine disorders) | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 1 | 0
PYREXIA (General disorders) | 2 | 0 | 1
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 0 | 1 | 0
BILE DUCT STONE (Hepatobiliary disorders) | 0 | 1 | 0
CHOLANGITIS (Hepatobiliary disorders) | 0 | 1 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 1 | 0
APPENDICITIS (Infections and infestations) | 0 | 1 | 0
ARTHRITIS INFECTIVE (Infections and infestations) | 0 | 0 | 1
ATYPICAL PNEUMONIA (Infections and infestations) | 1 | 0 | 0
BACTERIAL SEPSIS (Infections and infestations) | 0 | 0 | 1
CELLULITIS (Infections and infestations) | 1 | 0 | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 | 0 | 1
ENDOCARDITIS (Infections and infestations) | 1 | 1 | 0
ESCHERICHIA SEPSIS (Infections and infestations) | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 3 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
OSTEOMYELITIS (Infections and infestations) | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 3 | 2 | 3
POST PROCEDURAL INFECTION (Infections and infestations) | 0 | 1 | 0
PYELONEPHRITIS (Infections and infestations) | 0 | 1 | 1
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 | 1 | 0
SEPSIS (Infections and infestations) | 1 | 0 | 1
SINUSITIS (Infections and infestations) | 0 | 0 | 1
TOOTH INFECTION (Infections and infestations) | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 1 | 3
VIRAL INFECTION (Infections and infestations) | 1 | 0 | 0
ACUTE HAEMOLYTIC TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 | 1 | 0
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 | 1 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
COMA (Nervous system disorders) | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 1 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 | 1 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 0 | 0 | 1
SYNCOPE (Nervous system disorders) | 1 | 0 | 0
PRE-ECLAMPSIA (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
MAJOR DEPRESSION (Psychiatric disorders) | 0 | 0 | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 0 | 1
RENAL PAPILLARY NECROSIS (Renal and urinary disorders) | 1 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 0 | 0
ACUTE CHEST SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
STATUS ASTHMATICUS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
ABORTION INDUCED (Surgical and medical procedures) | 1 | 0 | 0
CENTRAL VENOUS CATHETERISATION (Surgical and medical procedures) | 0 | 1 | 0
HYSTERECTOMY (Surgical and medical procedures) | 1 | 0 | 0
ANGIOPATHY (Vascular disorders) | 0 | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 1
HYPOTENSION (Vascular disorders) | 1 | 0 | 0
VENOUS THROMBOSIS LIMB (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High-dose SelG1 (5.0 mg/kg SelG1) (N=66) | Low-dose SelG1 (2.5 mg/kg SelG10 (N=64) | Placebo (N=62)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 2 | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 | 3 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 4 | 0
CONSTIPATION (Gastrointestinal disorders) | 4 | 2 | 3
DIARRHOEA (Gastrointestinal disorders) | 7 | 5 | 1
NAUSEA (Gastrointestinal disorders) | 12 | 11 | 7
VOMITING (Gastrointestinal disorders) | 5 | 7 | 3
CHEST PAIN (General disorders) | 1 | 7 | 1
FATIGUE (General disorders) | 5 | 2 | 2
NON-CARDIAC CHEST PAIN (General disorders) | 3 | 2 | 4
PAIN (General disorders) | 2 | 3 | 6
PYREXIA (General disorders) | 5 | 6 | 3
NASOPHARYNGITIS (Infections and infestations) | 1 | 3 | 4
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 | 7 | 6
URINARY TRACT INFECTION (Infections and infestations) | 8 | 6 | 6
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 5 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 | 4 | 2
PROTHROMBIN TIME PROLONGED (Investigations) | 3 | 2 | 5
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 2 | 5
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 12 | 9 | 5
BACK PAIN (Musculoskeletal and connective tissue disorders) | 10 | 12 | 7
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 8 | 4 | 6
MYALGIA (Musculoskeletal and connective tissue disorders) | 5 | 2 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 11 | 8 | 10
DIZZINESS (Nervous system disorders) | 3 | 1 | 5
HEADACHE (Nervous system disorders) | 11 | 14 | 10
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 7
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 5 | 7 | 3

LIMITATIONS AND CAVEATS:
The Safety population includes all randomized patients who received at least one dose of study drug.

Although the safety is now coded with MedDRA 21.1, the CSR, when first published 1in 2016, used MedDRA 16.1 CFB = Change from Baseline

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.